CLINICAL TRIAL: NCT00222560
Title: The PAC Project: Integrating a Physical Activity Counsellor in the Primary Health Care Team: A Randomized Controlled Trial
Brief Title: The PAC Project: Integrating a Physical Activity Counsellor in the Primary Health Care Team
Acronym: PAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Hopital Montfort (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: G03-05441
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2007-04-30 (Estimated); Status verified 2007-04

CONDITIONS: Physical Inactivity
Keywords: physical activity counselling; physical activity behavior change intervention; prevention; collaborative health care; physical inactivity; motivation; fitness; randomized controlled trial
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Intensive physical activity counselling by an integrated physical activity counsellor

SUMMARY:
The Physical Activity Counselling (PAC) randomized controlled trial had as overall goal the establishment of a collaborative interdisciplinary primary care team to encourage physical activity. The main intervention was to integrate a physical activity counsellor to the primary care team so that the most appropriate care was given by the most appropriate provider. Much research has shown and many experts agree that patients need significant help to make and especially maintain physical activity behavior changes. Maintenance of these changes is essential for optimal health benefits. It was predicted that patients receiving both brief (2-4 minute) physical activity counselling from their family physician and intensive (3 month) physical activity counselling from an integrated physical activity counsellor (intensive counselling group) would report greater improvements in task motivation and task self-efficacy to engage in physical activity at the end of the intervention than those receiving only brief counselling (brief counselling group). The same was expected for both self-reported and objective physical activity. This RCT involved testing a theory-based counselling intervention, determining why the intervention was effective or ineffective by measuring key psychological mediating variables, using an objective measure to track changes in physical activity, and assessing physical and metabolic outcomes. This project represents an innovative theoretically based multi-level multi-intervention approach to promoting physical activity in primary care and is of great public health importance.

DETAILED DESCRIPTION:
Family doctors and nurses (health care providers - HCP) recommend that their patients are physically active because this is one of the most important things that patients can do to benefit their health. The Physical Activity Counselling (PAC) randomized controlled trial examined what happens when a physical activity counsellor is added to the family health care team. For the project, HCPs did a brief, 2-4 minute counselling session with their patients who reported doing less than 150 minutes of physical activity a week. Half (59) of the patients in the PAC Project only received this brief counselling from their HCP (brief counselling group) while the other half (61) also received six sessions with the physical activity counsellor over a three month period (intensive counselling group). The purpose of the project was to compare these 2 groups. The HCPs and the PAC used the 7 As shared-care model for physical activity counselling in primary care (Fortier et al., 2006). The HCPs and the PAC tried to help the patients want to (be motivated to) and to feel able to (be confident that they can) increase their level of physical activity. A number of validated questionnaires as well as some interviews were used to look at the effects of the counselling on motivation, confidence and physical activity. As well patients wore wear a small gadget known as an accelerometer to measure their actual physical activity. Quality of life was measured in all patients. Some patients (one third) had physical and metabolic testing three times during the trial. The cost of adding a PAC to a family health care team was also assessed.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 to 69 years
2. <150 minutes of physical activity/week
3. no uncontrolled medical conditions

Exclusion Criteria:

1. pregnancy (funder's request),
2. planned absence >3 weeks during the first 3 months of the study,
3. living with another patient in the study,
4. uncontrolled medical condition,
5. did not receive a physical activity prescription from their provider during the brief physical activity counselling,
6. received brief counselling more than once during the trial period and
7. uninterested in receiving intensive physical activity counselling

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-05; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
task motivation to engage in physical activity (0-100% motivated to engage in physical activity from 1-7 days a week in the next 6 weeks) | baseline, 6 weeks, 13 weeks, 19 weeks, 25 weeks
task self-efficacy to engage in physical activity (0-100% confident to engage in physical activity from 1-7 days a week in the next 6 weeks), measured every 6 weeks up to 25 weeks for maintenance | baseline, 6 weeks, 13 weeks, 19 weeks, 25 weeks

SECONDARY OUTCOMES:
Physical activity (subjective: in units with the Godin Leisure-Time Exercise Questionnaire) | baseline, 6 weeks, 13 weeks, 19 weeks, 25 weeks
physical activity (objective: in activity counts by the Actical accelerometer) | baseline, 13 weeks, 25 weeks
Quality of life | baseline, 13 weeks, 25 weeks
Physical and metabolic outcomes (33% sample) | baseline, 13 weeks, 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Fortier, PhD, Principal Investigator — University of Ottawa, Faculty of Health Sciences; William Hogg, MD, Principal Investigator — Department of Family Medicine, University of Ottawa and the C.T. Lamont Primary Health Care Research Centre, Élisabeth Bruyère Research Institute
Locations (1):
- Montfort Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Fortier M, Tulloch H, Hogg W. A good fit: integrating physical activity counselors into family practice. Can Fam Physician. 2006 Aug;52(8):942-4, 947-9. No abstract available. PMID 17273491
- [Background] Tulloch H, Fortier M, Hogg W. Physical activity counseling in primary care: who has and who should be counseling? Patient Educ Couns. 2006 Dec;64(1-3):6-20. doi: 10.1016/j.pec.2005.10.010. Epub 2006 Feb 10. PMID 16472959